CLINICAL TRIAL: NCT04829734
Title: Evaluation of the Effects of Photobiomodulation Therapy Combined With Static Magnetic Field (PBMT-sMF) on Temporary Pain Relief in Patients With Lateral Epicondylitis
Brief Title: Effects of Photobiomodulation Therapy Combined With Static Magnetic Field in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Multi Radiance Medical (Industry)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Principal investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.669.043
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Lateral Epicondylitis
Keywords: Photobiomodulation Therapy; Low-level Laser Therapy; Static Magnetic Fields; Epicondylitis; Intensity of Pain
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher will program the device (active PBMT-sMF or placebo PBMT-sMF) and will be instructed not to inform the patients or other researchers as to the type of treatment (active PBMT-sMF or placebo PBMT-sMF). Therefore, the researcher responsible for the treatment, the investigator and the outcome assessor will be blinded to the type of the treatment being administered to the patients. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active PBMT-sMF or placebo PBMT-sMF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active PBMT-sMF (Experimental): Active PBMT-sMF will be applied two times a week (three to four days apart), for three consecutive weeks, yielding six treatment sessions.
  Interventions: Device: Active PBMT-sMF
- Placebo PBMT-sMF (Placebo Comparator): Placebo PBMT-sMF will be applied two times a week (three to four days apart), for three consecutive weeks, yielding six treatment sessions.
  Interventions: Device: Placebo PBMT-sMF

INTERVENTIONS:
Device: Active PBMT-sMF — The Active PBMT-sMF will be applied using MRM® MR5 Prototype manufactured by Multi Radiance Medical (Solon, OH, USA). PBMT-sMF will be applied using the direct contact method with light pressure on the skin. The PBMT-sMF will be applied in four regions of the epicondyle and the application time will be 60 seconds per region. The total dose of PBMT-sMF will be 108,30 J per treatment session.
  Arms: Active PBMT-sMF
Device: Placebo PBMT-sMF — The Placebo PBMT-sMF will be applied using MRM® MR5 Prototype manufactured by Multi Radiance Medical (Solon, OH, USA). Placebo PBMT-sMF will be applied using the direct contact method with light pressure on the skin. The Placebo PBMT-sMF will be applied in four regions of the epicondyle and the application time will be 60 seconds per region. The total dose of Placebo PBMT-sMF will be 0 J per treatment session and the sMF will be turned off. The sounds and signals emitted from the device as well as the information displayed on the screen will be identical, regardless of the type of treatment (active or placebo).
  Arms: Placebo PBMT-sMF

SUMMARY:
Lateral epicondylitis (LE) is one of the most frequently encountered lesions affecting the upper extremity and is the most common cause of elbow pain in adults. It occurs on the lateral side of the elbow where the common extensors originate from the lateral epicondyle. LE can be considered an overuse injury which occurs on the lateral side of the elbow in the extensor tendons with repetitive micro-trauma. The clinical presentation of LE involves a painful or burning sensation over the humeral insertion of the common extensor tendons. Despite the high incidence of LE, optimal treatment has not been established. Treatment options include therapeutic exercise, bracing, shock wave or ultrasound therapy , but many of them lack sufficient evidence of beneficial effects. Photobiomodulation therapy (PBMT) alone or combined with static magnetic field (PBMT-sMF) has been shown to stimulate tendon healing, this suggests that therapy using laser or light-emitting diodes (LEDs) is efficacious for the symptoms associated with epicondylitis. According to the favorable results of PBMT-sMF in tendons repair processes, this type of therapy can be used as a therapeutic tool for management in epicondylitis, therefore, more investigations are necessary to establish the ideal parameters. Therefore, the aim of this project is to investigate the effects of PBMT-sMF, in the appropriate parameters, on degree of pain and quality of life of patients with lateral epicondylitis.

DETAILED DESCRIPTION:
To achieve the proposed objective it will be performed a multi-center, randomized, triple-blinded, placebo-controlled trial, with voluntary patients with lateral epicondylitis. Fifty patients will be randomly allocated to two treatment groups: 1. Active PBMT-sMF (MR5® Prototype Device) or Placebo PBMT-sMF (MR5® Prototype Device). The patients will be treated by a blinded therapist.

The patients randomly allocated to the different groups will be subjected to treatment two times a week for three consecutive weeks, each procedure administration three to four days apart.

The study will contain five phases: 1) pre-procedure activities; 2) pre-procedure assessment phase; 3) procedure administration phase; 4) procedure administration phase measures; 5) post-procedure administration phase.

The outcomes measured will be: degree of pain, forearm pain and disability, grip strength, TNF-α levels, subject satisfaction with overall outcome rating, perceived group assignment and adverse events.

The outcomes will be obtained at the stabilization phase (pre-procedure activities), baseline (pre-procedure assessment phase), 24 hours after the end of the treatment (procedure administration phase measures), and 30 days after the end of the treatment (post-procedure administration phase).

Statistical analysis:

1. The primary statistical method to analyze the primary endpoint will be Fisher's exact test to compare the proportion of success between the test (Active PBMT-sMF) and the control (Placebo PBMT-sMF) groups, considering that randomization has been diligently conducted and important covariates between the two groups are well balanced. Statistical significance will be set at p<0.05.
2. The secondary outcomes that are continuous variables will be analyzed through parametric analysis using ANCOVA. Statistical significance will be set at p<0.05.
3. For patient satisfaction, measured through a Likert Scale, the data will be reduced to the nominal level by combining all agree and disagree responses into two categories of "accept" and "reject". Differences in satisfaction with Study Outcome Ratings between procedure groups at both evaluated time-points, and any change between. The chi-square will be used after this transformation. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of pain around the lateral epicondyle for at least 1 month;
* Self-reported Degree of Pain rating on the 0-100 VAS pain scale for the lateral epicondyle region is 50 or greater;
* Tenderness localized to the epicondyle and anterodistal region of the epicondyle with palpation;
* 2 of 4 positive results of provocative tests comprising of Maudsley's, Cozen's, Thomsen and Mill's tests;
* Aged between 18 and 50 years;
* Both genders;
* Patients fluent in Portuguese.

Exclusion Criteria:

* hemophilia or any type of blood clotting disorder;
* chronic immune impairment neoplasia;
* cancer or treatment for cancer in the past 6 months, including tumors of the spinal cord;
* diabetes Type 1;
* significant heart conditions including CHF and implantable heart devices such as a pacemaker;
* current, active chronic pain disease: chronic fatigue syndrome, fibromyalgia, endometriosis, inflammatory bowel disease, interstitial cystitis diabetic neuropathic pain;
* neurologic deficits;
* cervical radiculopathy;
* peripheral nerve disease;
* rheumatoid arthritis;
* shoulder disease;
* radial tunnel syndrome;
* previous surgery of the affected upper extremities;
* congenital or acquired bony deformity in the ipsilateral upper extremity;
* bilateral epicondylosis;
* secondary orthopedic problems;
* the initiation of opioid analgesia or corticosteroid or analgesic injection interventions within the previous 6 months;
* local corticosteroids and/or botulinum toxin (Botox®) injection for Lateral Epicondyle pain relief within the prior 30 days;
* medical tx; such as chiropractic care and acupuncture within last 30 days;
* physical therapy intervention on the upper extremity in the previous year;
* active infection, wound, or other external trauma to the areas to be treated with the laser;
* medical, physical, or other contraindications for, or sensitivity to, light therapy;
* serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years;
* pregnant, breast feeding, or planning pregnancy prior to the end of study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] de Oliveira MFD, Leal-Junior ECP, Machado CDSM, Ribeiro NF, Dias LB, Lino MMA, Araujo-Silva OM, Casalechi HL, Johnson DS, Tomazoni SS. Effects of photobiomodulation therapy combined with static magnetic field on pain and function in patients with lateral epicondylitis: a multicentre, randomised, placebo-controlled trial. BMJ Open. 2025 Oct 5;15(10):e104789. doi: 10.1136/bmjopen-2025-104789. PMID 41047274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.64 (7.82) | 35.12 (9.77) | 34.88 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10 | 13 | 23
  Hispanic/Latino | 10 | 4 | 14
  African American | 4 | 8 | 12
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 25 | 25 | 50
Degree of pain rating (VAS) [Mean (Standard Deviation); unit: units on a scale] — Degree of pain rating was measured by 0-100 horizontal Visual Analog Pain Scale, with with 0 being 'no pain' and 100 'the worst possible pain'.
  units on a scale | 79.36 (10.19) | 75.60 (9.64) | 77.48 (10.00)
Forearm Pain and Disability [Mean (Standard Deviation); unit: units on a scale] — Were measured using the Patient-Rated Tennis Elbow Evaluation (PRTEE), which comprises 15 items divided into two subscales: a PAIN contained 5 questions about pain intensity (each item is rated from 0 = no pain and 10 = worst pain imaginable), and a FUCTION, contained 10 questions about how much difficulty the patient experiences when performing various daily or work-related tasks (each item is rated from 0 = no difficulty, 10 = inability to perform activities). These subscales are combined to yield a total score ranging from 0 to 100, with higher scores indicating greater impairment.
  units on a scale | 58.26 (9.45) | 59.28 (8.48) | 58.77 (8.90)
Grip Strength [Mean (Standard Deviation); unit: kgf] — The grip strength will be measured using a digital grip dynamometer type Jamar® Plus Digital Hand Dynamometer.
  kgf
    Affected/Treated Limb | 23.13 (8.16) | 24.24 (12.04) | 23.69 (10.19)
    Unaffected/ Untreated Limb | 24.71 (7.77) | 27.55 (12.46) | 26.13 (10.38)
TNF-α (Tumor Necrosis Factor-alpha) Levels [Mean (Standard Deviation); unit: pg/ml] — The TNF-α levels will be measured by blood samples through the enzyme-linked immunosorbent assay (ELISA).
  pg/ml | 35.75 (4.99) | 36.66 (6.96) | 36.20 (6.01)

OUTCOME MEASURES:

1. Primary Outcome: Degree of Pain Rating (VAS)
Description: Degree of pain rating will be measured by 0-100 horizontal Visual Analog Pain Scale, with with 0 being 'no pain' and 100 'the worst possible pain'
Time Frame: 3 weeks (end of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
units on a scale | 36.92 (22.64) | 51.40 (19.84)

2. Secondary Outcome: Forearm Pain and Disability
Description: Were measured using the Patient-Rated Tennis Elbow Evaluation (PRTEE), a 15-item questionnaire comprising five items related to pain and ten items related to function. Each item is rated on an 11-point scale ranging from 0 to 10, where 0 indicates no pain or difficulty and 10 indicates the worst imaginable pain or complete inability to perform the activity. The pain subscale score is obtained by summing the five pain items, yielding a maximum score of 50. The function subscale is calculated by summing the ten function items and dividing the total by 2, also resulting in a maximum score of 50. The total PRTEE score is the sum of the pain and function subscale scores, ranging from 0 (no pain or disability) to 100 (maximum pain and disability), with higher scores indicating greater impairment.
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
units on a scale
  Total scores - 3 weeks (end of treatment) | 39.44 (7.53) | 40.88 (8.61)
  Total scores - 4 weeks after the conclusion of the treatment | 29.60 (10.67) | 33.34 (9.68)
  Function scores - 3 weeks (end of treatment) | 14.28 (5.22) | 15.49 (8.61)
  Function scores - 4 weeks after the conclusion of the treatment | 10.72 (7.09) | 11.14 (6.36)

3. Secondary Outcome: Grip Strength
Description: The grip strength will be measured using a digital grip dynamometer type Jamar® Plus Digital Hand Dynamometer.
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Measure: Mean (Standard Deviation); unit: kgf
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
kgf
  3 weeks (end of treatment) - Affected/Treated Limb | 25.07 (8.83) | 26.37 (12.70)
  4 weeks after the conclusion of the treatment - Affected/Treated Limb | 25.97 (7.53) | 27.72 (12.60)
  3 weeks (end of treatment) - Unaffected/Untreated Limb | 25.45 (9.28) | 26.67 (12.57)
  4 weeks after the conclusion of the treatment - Unaffected/Untreated Limb | 26.07 (8.72) | 28.39 (11.23)

4. Secondary Outcome: TNF-α (Tumor Necrosis Factor-alpha) Levels
Description: The TNF-α levels will be measured by blood samples through the enzyme-linked immunosorbent assay (ELISA).
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
pg/ml
  3 weeks (end of treatment) | 25.77 (4.90) | 33.14 (4.71)
  4 weeks after the conclusion of the treatment | 26.45 (5.69) | 32.00 (6.11)

5. Secondary Outcome: Subject Satisfaction With Overall Outcome Rating
Description: Subject satisfaction will be measured by 1-item Likert Scale. The scale uses the following responses: 5 = Very Satisfied; 4 = Somewhat Satisfied; 3 = Neither Satisfied nor Dissatisfied; 2 = Not Very Satisfied; 1 = Not at All Satisfied. Highest scores indicates better satisfaction.
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
Participants
  3 weeks (end of treatment): Very satisfied | 18 | 16
  3 weeks (end of treatment): Somewhat Satisfied | 6 | 6
  3 weeks (end of treatment): Neither | 1 | 1
  3 weeks (end of treatment): Not Very Satisfied | 0 | 2
  3 weeks (end of treatment): Not at All Satisfied | 0 | 0
  4 weeks after the conclusion of the treatment: Very satisfied | 21 | 18
  4 weeks after the conclusion of the treatment: Somewhat Satisfied | 3 | 3
  4 weeks after the conclusion of the treatment: Neither | 1 | 3
  4 weeks after the conclusion of the treatment: Not Very Satisfied | 0 | 1
  4 weeks after the conclusion of the treatment: Not at All Satisfied | 0 | 0

6. Secondary Outcome: Presence of Adverse Events
Description: Adverse events will be measured by report.
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Measure: Number; unit: participants
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
participants
  Biting sensation | 1 | 0
  Heating of skin sensation | 1 | 0
  Pain and discomfort | 0 | 2
  Tingling sensation | 0 | 1

7. Secondary Outcome: Degree of Pain Rating (VAS)
Description: as for outcome 1
Time Frame: 4 weeks after the conclusion of the treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
Number analyzed (Participants) | 25 | 25
units on a scale | 20.28 (21.24) | 37.40 (24.08)

ADVERSE EVENTS:
Time Frame: 3 weeks (end of treatment) and 4 weeks after the conclusion of the treatment.
Arm/Group | Active PBMT-sMF | Placebo PBMT-sMF
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active PBMT-sMF (N=25) | Placebo PBMT-sMF (N=25)
Biting sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Heating (Skin and subcutaneous tissue disorders) | 1 (6) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Tingling sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT04829734/Prot_SAP_000.pdf